CLINICAL TRIAL: NCT05234281
Title: Concentrated Cross-disciplinary Group Intervention for Common Health Complaints (Mixed Anxiety Depression, Diabetes Mellitus Type 2, Low Back Pain, Chronic Obstructive Pulmonary Disease and Post COVID-19 Fatigue)
Brief Title: Concentrated Cross-disciplinary Group Intervention for Common Health Complaints (Including Post COVID-19 Fatigue)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helse i Hardanger (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020/101648
Record Dates: First submitted 2021-05-26; First posted 2022-02-10 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Mixed Anxiety Depression; Diabetes Mellitus, Type 2; Low Back Pain; Chronic Obstructive Pulmonary Disease; COVID-19
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Low Back Pain; Pulmonary Disease, Chronic Obstructive; COVID-19

STUDY DESIGN:
Intervention Model Description: Five groups of patients will be enrolled in this project, all in parallell, no randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low back pain (Other): Adults with chronic low back pain and at least 4 months of decreased work participation. Intervention as for all groups but with the use of GLADRyg back rehabilitation principles.
  Interventions: Other: Interdisciplincary concentrated group rehabilitation
- Chronic Obstructive Pulmonary Disease (COPD) (Other): Adults with COPD (FEV1<80%). Intervention as for all groups but with added pulmonary rehabilitation focus.
  Interventions: Other: Interdisciplincary concentrated group rehabilitation
- Diabetes type 2 (Other): Adults with type 2 diabetes and diabetes-related challenges including dysglycaemia, diabetic complications and/or weight issues. Intervention as for all groups but with added focus on how to make useful microchoices in terms of lifestyle.
  Interventions: Other: Interdisciplincary concentrated group rehabilitation
- Mixed anxiety/depression (Other): Young adults (18-35 years) with mixed anxiety/depression. Intervention as for all groups but with added focus on "acceptance and commitment therapy", behavioral analysis, metacognitive therapy and physical activity.
  Interventions: Other: Interdisciplincary concentrated group rehabilitation
- Post COVID-19 (Other): Adults who have persistant fatigue and/or dyspnea following infection with COVID-19.
  Interventions: Other: Interdisciplincary concentrated group rehabilitation

INTERVENTIONS:
Other: Interdisciplincary concentrated group rehabilitation — All arms receive a concentrated interdisciplinary rehabilitation with similar focus and structure:
  Three phases:
  1. Pre-intervention preparation (1-2 months): mobilize the patients' resources for change
  2. Concentrated group intervention (2-5 days): (further described below)
  3. Post-intervention follow-up (1 year): digital follow-up
  The core intervention is based on the concentrated rehabilitation format:
  1. Initiate treatment when the patient is ready for change
  2. Focus on the behavioral patterns which maintain the disorder, identify situations where they can break the patterns ("micro-choices").
  3. Assist the patient when breaking the patterns.
  4. Use long sessions to ensure that they face a broad range of potential micro-choices
  5. Work side-by side with others going through an analogous pattern of change
  6. Prepare them for taking responsibility for integrating the change into every-day living

SUMMARY:
The health care is faced by a growing challenge in the years to come: increasing age and chronic morbidity raising the costs, combined with decreased work participation. Among the conditions on the rise, we find anxiety/depression, musculoskeletal conditions, type 2 diabetes and chronic obstructive pulmonary disease. Recently, the rise of the Corona pandemic has yielded another group of (primarily young) patients with decreased work capacity, the post-Covid syndrome sufferers.

The aim of the present study is to establish, describe and summarize the experiences with a novel approach to rehabilitation for five of the most costly conditions; 1) low back pain, 2) chronic obstructive pulmonary disease, 3) type 2 diabetes mellitus, 4) mixed anxiety/depression and 5) post-Covid fatigue.

The concentrated interdisciplinary rehabilitation is characterised by three phases;

1. Pre-intervention preparation (1-2 months): with the aim to mobilize the patients' resources for change
2. Concentrated group intervention (2-5 days): interdisciplinary team - individually tailored training (further described below)
3. Post-intervention follow-up (1 year): digital follow-up with the aim of integrate the changes into everyday living

The concentrated intervention:

The core intervention is based on trans-diagnostic features of the highly successful 4-day intervention for Obsessive Compulsive Disorder, namely:

* Initiate treatment when the patient is ready for change
* Focus on the behavioral patterns which maintain the disorder and help the patient to identify situations where they can choose to break the pattern ("micro-choices").
* Assist the patient when they practice breaking the patterns. This may pertain to how they do physical training or to the way they walk, sit, eat, talk, take their medication and sleep, or to how they engage in social activities or take care of others.
* Use long sessions to ensure that they face a broad range of potential micro-choices
* Work side-by side with others going through an analogous pattern of change
* Prepare them for taking responsibility for integrating the change into every-day living

Main outcomes will be

1. Completion rates
2. Patient satisfaction
3. Changes to perception of illness
4. Patient activation

Secondary outcomes will be

1. Level of functioning
2. Qualitative description of participants' experiences

ELIGIBILITY:
Inclusion Criteria:

* Competent to consent
* Motivated to participate throughout the project
* Digital competence

Exclusion Criteria:

* Medical conditions that could preclude proper participation
* Unable to take care of everyday needs (nursing requirements)
* Cognitive failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Completion rates | 12 months
  Percentage of participants who are eligible for participation, who complete the 1 year programme
Patient satisfaction | 1 week post treatment and 12 months
  The Client Satisfaction Questionnaire (CSQ-8) is an 8-item questionnaire that measures patient satisfaction with health services, where the items are rated from 1 (very low satisfaction) to 4 (very high satisfaction). The total score ranges from 8-32, with higher scores indicating higher degree of satisfaction. The CSQ-8 has good psychometric properties, with high internal consistency (Cronbach's α = .93), and high inter-item correlation.
Changes to cognitive and emotional perception of illness | Baseline, 3, 6 and 12 months
  Changes (absolute levels and %) in cognitive and emotional representations of illness before, 3, 6 and 12 months after the intervention, as measured through the generic questionnaire The Brief Illness Perception Questionnaire (Brief IPQ). This is a 9-item questionnaire designed to assess cognitive and emotional representations of illness. Questions are graded from 1 to 10. The last item deals with perceived cause of illness, in which respondents list the perceived three most important causal factors in their illness. For this questionnaire, the general word 'illness' can be replaced by the name of a particular illness. The word 'treatment' in the treatment control item can be replaced by a particular treatment such as 'surgery' or 'physiotherapy'.
Changes in level of patient activation | Baseline, 3, 6 and 12 months
  Changes (absolute levels and %) in patient activation before, 3, 6 and 12 months after the intervention, as measured through the generic questionnaire Patient Activation Measure (PAM-13). This is the shortened version developed by Hibbard et al in 2005. Each question replied categorically as either disagree strongly, disagree, agree, agree strongly or N/A. These are further scored and summarized, yielding a 0-100 score, where higher score indicates higher degree of patient activation. The questionnaire is widely used, with high internal consistency (Cronbach's α = .91).

SECONDARY OUTCOMES:
Changes in level of functioning | Baseline, 3, 6 and 12 months
  Changes (absolute levels and %) in level of everyday function before, 3, 6 and 12 months after the intervention, as measured through the generic questionnaire Work and Social Adjustment Scale (WSAS). This short (6 item) questionnaire allows participants to grade their level of functioning on a 9-point scale, ranging from severly impaired to not impaired. The scale is widely used, and according to studies provide high internal consistencies ranging from Cronbach's α 0.70 to 0.94.

CONTACTS AND LOCATIONS:
Overall Officials: Eirik Søfteland, PhD, Principal Investigator — Helse i Hardanger
Locations (1):
- Helse i Hardanger, Øystese, Norway

REFERENCES:
- [Derived] Wilhelmsen-Langeland A, Bortveit T, Jurgensen M, Softeland E, Hystad SW, Kvale G. Concentrated transdiagnostic and cross-disciplinary micro-choice based group treatment for patients with depression and with anxiety leads to lasting improvements after 12 months: a pilot study. BMC Psychiatry. 2024 May 14;24(1):361. doi: 10.1186/s12888-024-05786-0. PMID 38745158
- [Derived] Kvale G, Softeland E, Jurgensen M, Wilhelmsen-Langeland A, Haugstvedt A, Hystad SW, Odegaard-Olsen OT, Aarli BB, Rykken S, Frisk B. First trans-diagnostic experiences with a novel micro-choice based concentrated group rehabilitation for patients with low back pain, long COVID, and type 2 diabetes: a pilot study. BMC Med. 2024 Jan 11;22(1):12. doi: 10.1186/s12916-023-03237-3. PMID 38200486
- [Derived] Frisk B, Njoten KL, Aarli B, Hystad SW, Rykken S, Kjosas A, Softeland E, Kvale G. A Novel Concentrated, Interdisciplinary Group Rehabilitation Program for Patients With Chronic Obstructive Pulmonary Disease: Protocol for a Nonrandomized Clinical Intervention Study. JMIR Res Protoc. 2022 Oct 26;11(10):e40700. doi: 10.2196/40700. PMID 36287602
- [Derived] Kvale G, Wilhelmsen-Langeland A, Jurgensen M, Hystad SW, Ost LG, Softeland E, Bortveit T. Concentrated transdiagnostic and cross-disciplinary group treatment for patients with depression and with anxiety: a pilot study. BMC Psychiatry. 2022 Sep 5;22(1):587. doi: 10.1186/s12888-022-04229-y. PMID 36058925

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT05234281/Prot_SAP_000.pdf